CLINICAL TRIAL: NCT04226976
Title: Efficacy of a Non-invasive Vestibular System Masking for the Abortive Treatment of Vertigo for Patients With Acute Unilateral Vestibulopathy (AUV)
Brief Title: Efficacy of a Non-invasive Vestibular System Masking for Improving Outcomes Following Acute Unilateral Vestibulopathy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 general concerns
Sponsor: Otolith Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLith10501
Record Dates: First submitted 2019-12-18; First posted 2020-01-13 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Dizziness; Nausea
MeSH Terms: conditions — Dizziness; Nausea

STUDY DESIGN:
Intervention Model Description: Participants with Acute Unilateral Vestibulopathy (AUV) will be asked to participate in the study. Subjects that give consent will be entered into the study and randomized to one of two groups (96dB or 98dB bone conduction level re:1dyne) by the study coordinator. Neither the subject nor the investigators in the study will know to which arm the subject was placed; rather the study coordinator will be given two sets of two OtoBands. When turned on, both the effective devices and placebo will be felt to vibrate, making it difficult for the typical subject or investigator to guess which device is effective and which is the placebo. After randomization, all subjects will undergo the vestibular battery. The subjects will complete a Participant Questionnaire following the testing.
Who Masked: Participant, Investigator
Masking Description: The sponsor will be randomly assigning the Otoband or placebo device to participants. The investigator will not know which device is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Otoband efficacy on AUV (Experimental): Participants will wear the Otoband during the single site visit against the skin, on the flat part of the right mastoid bone, about an inch behind the pinna and level with the ear canal. Half the participants will be given the Otoband at power level 96db and half will be given the Otoband at power level 98db (all bone conduction levels re:1dyne). This will be randomized and neither the participant nor the investigator will know what power level the Otoband is set at. The participants will be fitted with the Otoband and will undergo the vestibular battery test. The investigator will record the outcome measurements.
  Interventions: Device: Otoband
- Placebo device efficacy on AUV (Placebo Comparator): Participants will wear the placebo device during the single site visit against the skin, on the flat part of the right mastoid bone, about an inch behind the pinna and level with the ear canal. The placebo device will be set at a power level of 90db (bone conduction level re:1dyne). Neither the participant nor the investigator will know that this device is the placebo device. The participants will be fitted with the placebo device and will undergo the vestibular battery test. The investigator will record the outcome measurements.
  Interventions: Device: Placebo Device

INTERVENTIONS:
Device: Otoband — Participants with AUV will wear the Otoband set at normal power (effective) during vestibular test battery and outcome measurements will be recorded by the investigator during site visit.
  Arms: Otoband efficacy on AUV
Device: Placebo Device — Participants with AUV will wear the placebo device set at low power during vestibular test battery and outcome measurements will be recorded by the investigator during site visit.
  Arms: Placebo device efficacy on AUV

SUMMARY:
Vestibular disorders are among the most common causes of disability in society and affect over 50% of the population over the age of 65 and a significant percentage of the younger population. Acute unilateral vestibulopathy (AUV) is easy to diagnose and is commonly treated with physical therapy exercises called vestibular rehabilitation. But due to the discomfort experienced during AUV, patients can't usually comply with the treatment plan prescribed by their healthcare provider.

In this study, the investigators propose the use of an adjuvant device, the OtoBand, to improve balance, gait, reduce vertigo, and nausea in participants with AUV. Participants enrolled will undergo three vestibular tests batteries: one baseline, one with the OtoBand set at an effective power, and one with the placebo device set at low power. Neither participants nor investigator will know which device is effective and which is placebo. The OtoBand will be set at two different effective power levels. Which power level the participant will receive is randomized and unknown to the participant or investigator.

DETAILED DESCRIPTION:
Vestibular disorders are among the most common causes of disability in society and affect over 50% of the population over the age of 65 and a significant percentage of the younger population. Vestibular disorders have a dramatic impact on daily life impacting work, relationships, and even activities of daily living. At the current time, the mainstay of therapy for many vestibular disorders is a physical therapy called vestibular rehabilitation. While usually highly effective, this therapy is time consuming and not universally effective, in part because of inconsistent subject compliance. The use of adjuvant devices to speed recovery has been studied but very few devices have proved beneficial; the few that have shown benefit only work in special populations and are large units that cost several million dollars.

The OtoBand has shown promise and might be beneficial for treating or improving the course of recovery from vestibular disorders. To date, the device has only been systematically tested on healthy volunteers and has been shown to improve vertigo associated to motion sickness and virtual reality device use.

In this study, the investigators will assay the efficacy of the OtoBand on participants with acute unilateral vestibulopathy (AUV). The OtoBand will be given to participants with AUV for use during vestibular test batteries. The OtoBand will be set at either a normal power (effective) or low power (6 decibels lower than normal power, placebo device). There are two effective power levels, which will be randomly assigned to each of the participants. Outcomes will be assessed by the investigator by a set of vestibular tests while the participant uses the OtoBand or placebo device. Participants vestibular disorder outcomes will be compared between OtoBand and placebo device to:

1. Determine if participants treated with OtoBand achieve instantaneous effectiveness in reducing vestibular symptoms.
2. Determine if participants treated with the OtoBand at higher power levels experience higher benefits.

ELIGIBILITY:
Inclusion Criteria:

Subject between the ages of 18-70 with an acute unilateral vestibulopathy as characterized by the following

* Acute onset vertigo that lasts at least 6 hours within the previous 2 weeks.
* A feeling of unsteadiness or feeling off balance for at least 48 hours after conclusion of vertigo
* Confirmed unilateral vestibulopathy on head rotation test or caloric test

Exclusion Criteria:

1. Resolved vestibular hypofunction by the time of visit to clinic
2. History of head injury within the last six months or currently suffering the effects of a head injury
3. Presence of severe aphasia
4. History of diagnosed, untreated neuropsychiatric disorders (e.g. hypochondriasis, major depression, schizophrenia)
5. Documented neurodegenerative disorders
6. Prior disorders of hearing and balance including:

   1. Ménière's disease
   2. Multiple sclerosis
   3. Vestibular neuritis (prior resolved episode)
   4. Vestibular schwannoma
   5. Sudden sensorineural hearing loss
7. History of Cerebrovascular disorders
8. History of ear operation other than myringotomy (tube placement) in the past
9. Systemic disorders to include chronic renal failure, cirrhosis of the liver, autoimmune disease, heart disease, lung disease, or severe arthritis
10. Individuals who cannot provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in vestibular function as measured by Functional Gait Assessment | Three tests over 30 minutes - During 1-day visit at the University of Miami Health System.
  Measure statistically significant change in postural stability in acute vestibular patients, by obtaining the participants' scores on the Functional Gait Assessment (FGA). An ANOVA will be performed on the FGA scores - without a device, - with an Otoband set at a subtherapeutic power level and - with an Otoband set at a therapeutic power level.
Change in vestibular function as measured by Dizziness Handicap Inventory | Three times immediately following FGA testing - During 1-day visit at the University of Miami Health System.
  Measure statistically significant change in perception of dizziness by administering the Dizziness Handicap Inventory (DHI) immediately following the gait tasks of the Functional Gait Assessment. An ANOVA comparison will be performed between the set of DHI scores - without a device, - with an Otoband set at a subtherapeutic power level and - with an Otoband set at a therapeutic power level.
Change in vestibular function as measured by I-PAS testing | Three tests over one hour - During the 1-day visit at the University of Miami Health System.
  Measure statistically significant change in vestibular function and reduction in vestibular symptoms, as measured from the participant's score on the I-PAS test battery. The I-PAS consists in "video Head Impulse Testing" (vHIT) and the "Oculomotor, Vestibular, and Reaction Time" testing (OVRT). An ANOVA comparison will be performed between the set of scoresI-PAS scores - without a device, - with an Otoband set at a subtherapeutic power level and - with an Otoband set at a therapeutic power level.

SECONDARY OUTCOMES:
Differential effect of bone conduction level on vestibular improvements | Summary data at end of study (1 year)
  The trial has two groups of participants: half of the participants are tested with the OtoBand set at a bone conduction level found to be optimally effective in healthy subjects, and half of the participants are tested with the OtoBand set at a higher bone conduction level. A statistical test will be used to determine whether acute unilateral vestibulopathy participants, as a group, experience higher or lower benefits from the higher bone conduction power level, using the measures of the three primary outcomes (FGA, DHI, I-PAS).

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Study Director — Otolith Labs
Locations (1):
- University of Miami Health System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No